CLINICAL TRIAL: NCT02246998
Title: A Randomized, Open Label, Phase 4 Study Evaluating the Renal Effect of Elvitegravir/Cobicistat/Emtricitabine/Tenofovir DF or Other Tenofovir DF-containing Regimens (Ritonavir-boosted Atazanavir Plus Emtricitabine/Tenofovir DF or Efavirenz/Emtricitabine/Tenofovir DF) Compared to Ritonavir-boosted Atazanavir Plus Abacavir/Lamivudine in Antiretroviral Treatment-naïve HIV-1 Infected Adults With eGFR ≥70 mL/Min
Brief Title: Renal Effect of Stribild or Other Tenofovir DF-containing Regimens Compared to Ritonavir-boosted Atazanavir Plus Abacavir/Lamivudine in Antiretroviral Treatment-naive HIV-1 Infected Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-236-0140; 2014-002095-93 (EudraCT Number)
Record Dates: First submitted 2014-09-19; First posted 2014-09-23 (Estimated); Results first posted 2018-01-03 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Ritonavir; Atazanavir Sulfate; abacavir, lamivudine drug combination; Iohexol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- STB+iohexol (Experimental): Participants will receive STB+iohexol for 24 weeks.
  Interventions: Drug: STB; Drug: Iohexol
- RTV+ATV+TVD+iohexol (Experimental): Participants will receive RTV+ATV+TVD+iohexol for 24 weeks.
  Interventions: Drug: TVD; Drug: RTV; Drug: ATV; Drug: Iohexol
- ATR+iohexol (Experimental): Participants will receive ATR+iohexol for 24 weeks.
  Interventions: Drug: ATR; Drug: Iohexol
- RTV+ATV+ABC/3TC+iohexol (Experimental): Participants will receive RTV+ATV+ABC/3TC+iohexol for 24 weeks.
  Interventions: Drug: RTV; Drug: ATV; Drug: ABC/3TC; Drug: Iohexol

INTERVENTIONS:
Drug: STB — 150/150/200/300 mg fixed dose combination (FDC) tablet administered orally once daily with food
  Other Names: Stribild®
  Arms: STB+iohexol
Drug: TVD — 200/300 mg FDC tablet administered orally once daily with food
  Other Names: Truvada®
  Arms: RTV+ATV+TVD+iohexol
Drug: ATR — 600/200/300 mg FDC tablet administered orally once daily on an empty stomach at bedtime
  Other Names: Atripla®
  Arms: ATR+iohexol
Drug: RTV — 100 mg tablet administered orally once daily with food
  Other Names: Norvir®
  Arms: RTV+ATV+ABC/3TC+iohexol; RTV+ATV+TVD+iohexol
Drug: ATV — 300 mg capsule administered orally once daily with food
  Other Names: Reyataz®
  Arms: RTV+ATV+ABC/3TC+iohexol; RTV+ATV+TVD+iohexol
Drug: ABC/3TC — 600/300 mg FDC tablet administered orally once daily with food
  Other Names: Kivexa®
  Arms: RTV+ATV+ABC/3TC+iohexol
Drug: Iohexol — 1500 mg solution administered intravenously at baseline, and at Weeks 4, 8, 16, and 24
  Other Names: Omnipaque™

SUMMARY:
The primary objective of this study is to assess glomerular function before and during administration of stribild (STB; elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate (E/C/F/TDF)) or a regimen containing TDF without cobicistat (COBI) as ritonavir (RTV)-boosted atazanavir (ATV/r) plus truvada (TVD; FTC/TDF) or atripla (ATR; efavirenz/emtricitabine/tenofovir disoproxil fumarate (EFV/FTC/TDF)) compared to a regimen containing neither TDF nor COBI as ATV/r plus abacavir/lamivudine (ABC/3TC) via determination of actual glomerular filtration rate (aGFR) using iohexol (a probe GFR marker) plasma clearance and estimated (calculated) glomerular filtration rate (eGFR).

ELIGIBILITY:
Key Inclusion Criteria:

* Treatment naïve
* Plasma HIV-1 RNA levels ≥ 5,000 copies/mL at Screening
* CD4 cell count > 200 cells/µL
* Screening genotype report provided by the site must show sensitivity to FTC, TDF, EFV, ABC, 3TC, ATV and absence of study drug resistance mutations that include K65R, K70E and M184V in RT
* Estimated GFR ≥ 70 mL/min
* Hepatic transaminases (aspartate aminotransferase [AST] and alanine aminotransferase [ALT]) ≤ 5 × upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 mg/dL (≤ 26 umol/L), or normal direct bilirubin
* Adequate hematologic function (absolute neutrophil count ≥ 1,000/mm^3; platelets ≥ 50,000/mm^3; hemoglobin ≥ 8.5 g/dL)
* Serum amylase ≤ 5 × ULN (individuals with serum amylase > 5 × ULN will remain eligible if serum lipase is ≤ 5 × ULN)
* Normal electrocardiogram (ECG) or not clinically significant if abnormal ECG
* Not pregnant or non-lactating females of non-childbearing potential. Or females with childbearing potential who agree to utilize highly effective contraception methods or be non-heterosexually active or practice sexual abstinence from screening throughout the duration of study treatment and for 90 days if taking EFV/FTC/TDF or for 30 days for all other study drugs following the last study drug dose
* Males who agree to utilize a highly effective method of contraception during heterosexual intercourse or be non-heterosexually active, or practice sexual abstinence from first dose throughout the study period and for 90 days if taking EFV/FTC/TDF or for 30 days for all other study drugs following the last study drug dose. Males who agree to refrain from sperm donation from first dose until at least 90 days if taking EFV/FTC/TDF or for 30 days for all other study drugs following the last study drug dose
* Body mass index (BMI) of 19 ≤ BMI ≤ 30 kg/m^2 and body weight ≥ 40 kg
* Life expectancy ≥ 1 year

Key Exclusion Criteria:

* HLA-B*5701 allele positive
* A new AIDS-defining condition diagnosed within the 30 days prior to screening
* Hepatitis B surface antigen (HBsAg) positive
* Hepatitis C virus (HCV) antibody positive and HCV RNA detectable
* Individuals experiencing decompensated cirrhosis
* Females who are breastfeeding
* Positive serum pregnancy test
* Have an implanted defibrillator or pacemaker
* Current alcohol or substance that could potentially interfere with study compliance
* A history of malignancy within the past 5 years (prior to screening) or ongoing malignancy other than cutaneous Kaposi's sarcoma (KS), basal cell carcinoma, or resected, non-invasive cutaneous squamous carcinoma. Individuals with cutaneous KS are eligible, but must not have received any systemic therapy for KS within 30 days of Day 1 Visit and must not be anticipated to require systemic therapy during the study
* Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to Day 1 Visit

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2014-12-15 (Actual); Primary Completion 2016-01-20 (Actual); Study Completion 2016-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (20):
- Belgium (2):
  - Brussels
  - Ghent
- France (4):
  - Lyon
  - Paris
  - Rennes
  - Tourcoing
- Dublin, Ireland
- Spain (3):
  - Barcelona
  - Madrid
  - Seville
- United Kingdom (10):
  - Birmingham
  - Bournemouth
  - Brighton
  - Bristol
  - Coventry
  - Liverpool
  - London
  - Manchester
  - Newcastle
  - Sheffield

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Belgium, Ireland, Spain, and the United Kingdom. The first participant was screened on 15 Dec 2014. The last study visit occurred on 17 February 2016.
Pre-assignment Details: 93 participants were screened.
Groups:
- STB + Iohexol: Elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate (STB; Stribild®; EVG/COBI/FTC/TDF; 150/150/200/300 mg) FDC tablet orally with food once daily for 24 weeks + iohexol 1500 mg solution administered intravenously at Baseline (Day1), and Weeks 4, 8, 16, and 24
- TVD + ATV/r + Iohexol: FTC/TDF (TVD; Truvada®; 200/300 mg) FDC tablet + Atazanavir (ATV) 300 mg capsule + Ritonavir (RTV) 100 mg tablet orally with food once daily for 24 weeks + iohexol 1500 mg solution administered intravenously at Baseline (Day 1), and Weeks 4, 8, 16, and 24
- ATR + Iohexol: EFV/FTC/TDF (ATR; Atripla® 600/200/300 mg) FDC tablet orally once daily on an empty stomach for 24 weeks + iohexol 1500 mg solution administered intravenously at Baseline (Day1), and Weeks 4, 8, 16, and 24
- ABC/3TC + ATV/r + Iohexol: ABC/3TC (600/300 mg) FDC tablet + ATV 300 mg capsule + RTV 100 mg tablet orally with food once daily for 24 weeks + iohexol 1500 mg solution administered intravenously at Baseline (Day1), and Weeks 4, 8, 16, and 24
Period: Overall Study
Arm/Group | STB + Iohexol | TVD + ATV/r + Iohexol | ATR + Iohexol | ABC/3TC + ATV/r + Iohexol
Started | 18 | 18 | 18 | 18
Completed | 16 | 15 | 15 | 16
Not Completed | 2 | 3 | 3 | 2
Not completed — Adverse Event | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1
Not completed — Randomized but Never Dosed | 1 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: all randomized participants who received at least 1 dose of study drug, excluding iohexol
Groups:
- STB + Iohexol: STB (150/150/200/300 mg) FDC tablet orally with food once daily for 24 weeks + iohexol 1500 mg solution administered intravenously at Baseline (Day1), and Weeks 4, 8, 16, and 24
- TVD + ATV/r + Iohexol: TVD (200/300 mg) FDC tablet + ATV 300 mg capsule + RTV 100 mg tablet orally with food once daily for 24 weeks + iohexol 1500 mg solution administered intravenously at Baseline (Day 1), and Weeks 4, 8, 16, and 24
- ATR + Iohexol: ATR (600/200/300 mg) FDC tablet orally once daily on an empty stomach for 24 weeks + iohexol 1500 mg solution administered intravenously at Baseline (Day1), and Weeks 4, 8, 16, and 24
- Total: Total of all reporting groups
Arm/Group | STB + Iohexol | TVD + ATV/r + Iohexol | ATR + Iohexol | ABC/3TC + ATV/r + Iohexol | Total
Number analyzed (Participants) | 17 | 16 | 16 | 17 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (8.1) | 34 (8.4) | 34 (9.6) | 34 (7.5) | 35 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 0 | 2
  Male | 17 | 15 | 15 | 17 | 64
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 1 | 2
  Black | 2 | 1 | 2 | 1 | 6
  White | 13 | 15 | 13 | 15 | 56
  Other | 0 | 0 | 1 | 0 | 1
  Hispanic or Latino | 2 | 3 | 2 | 0 | 7
  Not Hispanic or Latino | 15 | 13 | 14 | 17 | 59
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 3 | 2 | 5 | 4 | 14
  Ireland | 1 | 3 | 1 | 0 | 5
  United Kingdom | 11 | 9 | 9 | 8 | 37
  Spain | 3 | 4 | 3 | 6 | 16
Actual Glomerular Filtration Rate [Mean (Standard Deviation); unit: mL/min] | 111.8 (31.07) | 112.0 (19.17) | 105.4 (38.22) | 96.6 (34.52) | 106.4 (31.52)
Estimated Glomerular Filtration Rate by Cockcroft-Gault [Mean (Standard Deviation); unit: mL/min] | 120.8 (13.94) | 121.2 (24.34) | 119.5 (20.36) | 122.6 (20.25) | 121.0 (19.55)
Estimated Glomerular Filtration Rate by MDRD Formula [Mean (Standard Deviation); unit: mL/min/1.73m2] | 103.8 (14.06) | 110.6 (18.47) | 108.4 (21.42) | 105.5 (12.59) | 107.0 (16.71)
CD4 Cell Count [Mean (Standard Deviation); unit: cells/uL] | 552 (177.8) | 600 (217.9) | 553 (215.8) | 524 (190.0) | 557 (197.8)

OUTCOME MEASURES:

1. Primary Outcome: Actual Glomerular Filtration Rate (aGFR) Using Iohexol Plasma Clearance (CLiohexol) at Week 24
Time Frame: Week 24
Population: Participants in the pharmacodynamics (PD) analysis Set (all treated participants in each group, who have evaluable baseline and at least 1 postbaseline aGFR and /or eGFR at any visit) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | STB + Iohexol | TVD + ATV/r + Iohexol | ATR + Iohexol | ABC/3TC + ATV/r + Iohexol
Number analyzed (Participants) | 17 | 15 | 15 | 17
mL/min | 103.6 (23.28) | 104.9 (27.16) | 111.1 (23.23) | 101.0 (27.01)

2. Primary Outcome: Estimated GFR (eGFR) Calculated by Cockcroft-Gault Formula at Week 24
Description: GFR is a measure of the rate at which blood is filtered by the kidney. Cockcroft-Gault is an equation (calculation) used to estimate GFR based on serum creatinine, weight, and gender. eGFR = (140 - age) * (mass in kg) * (0.85 if female) divided by 72 * serum creatinine in mg/dL
Time Frame: Week 24
Population: Participants in the PD Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | STB + Iohexol | TVD + ATV/r + Iohexol | ATR + Iohexol | ABC/3TC + ATV/r + Iohexol
Number analyzed (Participants) | 16 | 15 | 15 | 16
mL/min | 116.9 (17.06) | 122.4 (31.71) | 120.0 (20.52) | 123.0 (25.74)

3. Primary Outcome: Estimated GFR Calculated by Modification of Diet in Renal Disease (MDRD) Formula at Week 24
Description: MDRD is an equation (calculation) used to estimate GFR in participants with impaired renal function based on serum creatinine, age, race, and gender. eGFR (mL/min/1.73 m^2) = 186 * (Scr)^-1.154 * (Age)^(-0.203) * (0.742 if female) * (1.212 if black). Scr = serum creatinine in mg/dL
Time Frame: Week 24
Population: Participants in the PD Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | STB + Iohexol | TVD + ATV/r + Iohexol | ATR + Iohexol | ABC/3TC + ATV/r + Iohexol
Number analyzed (Participants) | 16 | 15 | 15 | 16
mL/min/1.73m^2 | 99.3 (17.07) | 110.2 (23.98) | 109.2 (20.90) | 104.9 (12.59)

4. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Graded Laboratory Abnormality: Urine Glucose (by Dipstick)
Time Frame: Up to 24 weeks plus 30 days
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | STB + Iohexol | TVD + ATV/r + Iohexol | ATR + Iohexol | ABC/3TC + ATV/r + Iohexol
Number analyzed (Participants) | 17 | 16 | 16 | 17
Participants
  Grade 1 | 0 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0
  Any Grade | 0 | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Graded Laboratory Abnormality: Serum Glucose (Fasting)
Time Frame: Up to 24 weeks plus 30 days
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | STB + Iohexol | TVD + ATV/r + Iohexol | ATR + Iohexol | ABC/3TC + ATV/r + Iohexol
Number analyzed (Participants) | 17 | 16 | 15 | 17
percentage of participants
  Grade 1 (Hyperglycemia) | 11.8 | 12.5 | 20.0 | 0
  Grade 1 (Hypoglycemia) | 0 | 0 | 0 | 0
  Grade 2 (Hyperglycemia) | 0 | 0 | 0 | 0
  Grade 2 (Hypoglycemia) | 0 | 6.3 | 0 | 0
  Grade 3 (Hyperglycemia) | 0 | 0 | 0 | 0
  Grade 3 (Hypoglycemia) | 0 | 0 | 0 | 0
  Grade 4 (Hyperglycemia) | 0 | 0 | 0 | 0
  Grade 4 (Hypoglycemia) | 0 | 0 | 0 | 0
  Any grade (Hyperglycemia) | 11.8 | 12.5 | 20.0 | 0
  Any grade (Hypoglycemia) | 0 | 6.3 | 0 | 0

6. Secondary Outcome: Percentage Change From Baseline in Urine Albumin to Creatinine Ratio (mg/g) at Week 24
Time Frame: Baseline; Week 24
Population: Participants in the PD Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | STB + Iohexol | TVD + ATV/r + Iohexol | ATR + Iohexol | ABC/3TC + ATV/r + Iohexol
Number analyzed (Participants) | 16 | 14 | 13 | 17
percentage change | 0.0 [-23.6 to 50.0] | -18.3 [-57.1 to 50.0] | 50.0 [-25.0 to 100.0] | -16.7 [-37.5 to 0.0]

7. Secondary Outcome: Percentage Change From Baseline in Urine Protein to Creatinine Ratio (mg/g) at Week 24
Time Frame: Baseline; Week 24
Population: Participants in the PD Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | STB + Iohexol | TVD + ATV/r + Iohexol | ATR + Iohexol | ABC/3TC + ATV/r + Iohexol
Number analyzed (Participants) | 16 | 14 | 15 | 17
percentage change | 5.7 [-11.0 to 22.5] | 17.5 [0.0 to 45.7] | -10.5 [-41.9 to 69.8] | 7.1 [-24.3 to 13.3]

8. Secondary Outcome: Percentage Change From Baseline in Urine β2-microglobulin to Creatinine Ratio (µg/g) at Week 24
Time Frame: Baseline; Week 24
Population: Participants in the PD Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | STB + Iohexol | TVD + ATV/r + Iohexol | ATR + Iohexol | ABC/3TC + ATV/r + Iohexol
Number analyzed (Participants) | 16 | 14 | 13 | 17
percentage change | -5.1 [-48.2 to 22.8] | 197.3 [21.7 to 328.7] | -1.1 [-33.1 to 36.7] | -22.7 [-60.8 to -6.0]

9. Secondary Outcome: Percentage Change From Baseline in Urine Retinol Binding Protein (RBP) to Creatinine Ratio (µg/g) at Week 24
Time Frame: Baseline; Week 24
Population: Participants in the PD Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | STB + Iohexol | TVD + ATV/r + Iohexol | ATR + Iohexol | ABC/3TC + ATV/r + Iohexol
Number analyzed (Participants) | 16 | 14 | 13 | 17
percentage change | 38.1 [-1.1 to 51.1] | 52.2 [5.9 to 147.6] | 52.1 [-33.8 to 92.8] | 4.8 [-13.6 to 15.5]

10. Secondary Outcome: Pharmacokinetic (PK) Parameter: Cmax for COBI
Description: Cmax is defined as the maximum observed concentration of drug in plasma.
Time Frame: Pre-dose, 0, 0.5, 1, 2, 3, 4, 5, 6, and 10 hours post "time zero" at Weeks 4, 8, 16, and 24
Population: Participants in the COBI PK Analysis Set (all treated participants who have respective, evaluable PK profiles of COBI) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | STB + Iohexol
Number analyzed (Participants) | 17
ng/mL
  Week 4 | 1189.1 (377.88)
  Week 8 | 1017.8 (388.09)
  Week 16 | 1197.3 (656.33)
  Week 24: number analyzed (Participants) | 16
  Week 24 | 1123.4 (430.41)

11. Secondary Outcome: PK Parameter: Tmax for COBI
Description: Tmax is defined as the time of Cmax.
Time Frame: Pre-dose, 0, 0.5, 1, 2, 3, 4, 5, 6, and 10 hours post "time zero" at Weeks 4, 8, 16, and 24
Population: Participants in the COBI PK Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | STB + Iohexol
Number analyzed (Participants) | 17
hours
  Week 4 | 3.3 [3.0 to 4.1]
  Week 8 | 3.1 [3.0 to 4.1]
  Week 16 | 3.1 [2.1 to 4.0]
  Week 24: number analyzed (Participants) | 16
  Week 24 | 3.0 [2.1 to 4.0]

12. Secondary Outcome: PK Parameter: Clast for COBI
Description: Clast is defined as the last observable concentration of drug.
Time Frame: Pre-dose, 0, 0.5, 1, 2, 3, 4, 5, 6, and 10 hours post "time zero" at Weeks 4, 8, 16, and 24
Population: Participants in the COBI PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | STB + Iohexol
Number analyzed (Participants) | 17
ng/mL
  Week 4 | 85.0 (126.69)
  Week 8 | 54.5 (59.58)
  Week 16 | 214.0 (693.66)
  Week 24: number analyzed (Participants) | 16
  Week 24 | 162.7 (299.48)

13. Secondary Outcome: PK Parameter: Tlast for COBI
Description: * Tlast is defined as the time of Clast.
  * Plasma samples for PK analysis were collected out to 10 hours postdose, and the predose concentration was used as a surrogate for the 24 hour concentration for PK parameter generation.
Time Frame: Pre-dose, 0, 0.5, 1, 2, 3, 4, 5, 6, and 10 hours post "time zero" at Weeks 4, 8, 16, and 24
Population: Participants in the COBI PK Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | STB + Iohexol
Number analyzed (Participants) | 17
hours
  Week 4 | 24.0 [24.0 to 24.0]
  Week 8 | 24.0 [24.0 to 24.0]
  Week 16 | 24.0 [24.0 to 24.0]
  Week 24: number analyzed (Participants) | 16
  Week 24 | 24.0 [10.1 to 24.0]

14. Secondary Outcome: PK Parameter: Ctau for COBI
Description: Ctau is defined as the observed drug concentration at the end of the dosing interval.
Time Frame: Pre-dose, 0, 0.5, 1, 2, 3, 4, 5, 6, and 10 hours post "time zero" at Weeks 4, 8, 16, and 24
Population: Participants in the COBI PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | STB + Iohexol
Number analyzed (Participants) | 17
ng/mL
  Week 4 | 59.7 (113.31)
  Week 8 | 26.0 (28.79)
  Week 16 | 198.3 (697.06)
  Week 24 | 82.7 (285.81)

15. Secondary Outcome: PK Parameter: λz for COBI
Description: λz is defined as the terminal elimination rate constant.
Time Frame: Pre-dose, 0, 0.5, 1, 2, 3, 4, 5, 6, and 10 hours post "time zero" at Weeks 4, 8, 16, and 24
Population: Participants in the COBI PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | STB + Iohexol
Number analyzed (Participants) | 16
1/hour
  Week 4 | 0.179 (0.0598)
  Week 8: number analyzed (Participants) | 15
  Week 8 | 0.192 (0.0481)
  Week 16 | 0.206 (0.0610)
  Week 24: number analyzed (Participants) | 15
  Week 24 | 0.211 (0.0844)

16. Secondary Outcome: PK Parameter: AUCtau for COBI
Description: AUCtau is defined as the concentration of drug over time (area under the plasma concentration versus time curve over the dosing interval).
Time Frame: Pre-dose, 0, 0.5, 1, 2, 3, 4, 5, 6, and 10 hours post "time zero" at Weeks 4, 8, 16, and 24
Population: Participants in the COBI PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | STB + Iohexol
Number analyzed (Participants) | 17
h*ng/mL
  Week 4: number analyzed (Participants) | 16
  Week 4 | 9225.8 (2786.60)
  Week 8: number analyzed (Participants) | 15
  Week 8 | 8127.4 (3217.12)
  Week 16 | 10684.8 (12567.09)
  Week 24: number analyzed (Participants) | 15
  Week 24 | 8391.3 (6132.50)

17. Secondary Outcome: PK Parameter: t1/2 for COBI
Description: t1/2 is defined as the estimate of the terminal elimination half-life of the drug.
Time Frame: Predose, 0, 0.5, 1, 2, 3, 4, 5, 6, and 10 hours post "time zero" at Weeks 4, 8, 16, and 24
Population: Participants in the COBI PK Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | STB + Iohexol
Number analyzed (Participants) | 17
hours
  Week 4: number analyzed (Participants) | 16
  Week 4 | 3.80 [3.24 to 4.63]
  Week 8: number analyzed (Participants) | 15
  Week 8 | 4.09 [2.89 to 4.75]
  Week 16: number analyzed (Participants) | 16
  Week 16 | 3.42 [2.91 to 4.18]
  Week 24: number analyzed (Participants) | 15
  Week 24 | 3.24 [2.57 to 4.39]

18. Secondary Outcome: PK Parameter: Cmax for RTV
Time Frame: Pre-dose, 0, 0.5, 1, 2, 3, 4, 5, 6, and 10 hours post "time zero" at Weeks 4, 8, 16, and 24
Population: Participants in the RTV PK Analysis Set (all treated participants who have respective, evaluable PK profiles of RTV) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TVD + ATV/r + Iohexol | ABC/3TC + ATV/r + Iohexol
Number analyzed (Participants) | 16 | 17
ng/mL
  Week 4 | 1260.0 (453.58) | 1352.1 (513.74)
  Week 8 | 1142.3 (489.18) | 1326.2 (493.47)
  Week 16: number analyzed (Participants) | 15 | 17
  Week 16 | 1144.8 (416.41) | 1557.6 (555.87)
  Week 24: number analyzed (Participants) | 15 | 17
  Week 24 | 1217.7 (445.18) | 1485.4 (662.49)

19. Secondary Outcome: PK Parameter: Tmax for RTV
Time Frame: Pre-dose, 0, 0.5, 1, 2, 3, 4, 5, 6, and 10 hours post "time zero" at Weeks 4, 8, 16, and 24
Population: Participants in the RTV PK Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | TVD + ATV/r + Iohexol | ABC/3TC + ATV/r + Iohexol
Number analyzed (Participants) | 16 | 17
hours
  Week 4 | 4.0 [3.2 to 4.6] | 4.0 [2.1 to 4.1]
  Week 8 | 4.0 [2.5 to 5.1] | 4.0 [3.0 to 4.1]
  Week 16: number analyzed (Participants) | 15 | 17
  Week 16 | 4.1 [3.0 to 5.1] | 4.0 [2.2 to 4.1]
  Week 24: number analyzed (Participants) | 15 | 17
  Week 24 | 4.0 [3.0 to 5.0] | 4.0 [3.0 to 4.1]

20. Secondary Outcome: PK Parameter: Clast for RTV
Time Frame: Pre-dose, 0, 0.5, 1, 2, 3, 4, 5, 6, and 10 hours post "time zero" at Weeks 4, 8, 16, and 24
Population: Participants in the RTV PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TVD + ATV/r + Iohexol | ABC/3TC + ATV/r + Iohexol
Number analyzed (Participants) | 16 | 17
ng/mL
  Week 4 | 59.5 (57.85) | 61.0 (56.51)
  Week 8 | 71.0 (91.24) | 85.5 (99.68)
  Week 16: number analyzed (Participants) | 15 | 17
  Week 16 | 69.2 (49.85) | 99.1 (92.42)
  Week 24: number analyzed (Participants) | 15 | 17
  Week 24 | 102.5 (182.16) | 187.9 (258.53)

21. Secondary Outcome: PK Parameter: Tlast for RTV
Description: Plasma samples for PK analysis were collected out to 10 hours postdose, and the predose concentration was used as a surrogate for the 24 hour concentration for PK parameter generation.
Time Frame: Pre-dose, 0, 0.5, 1, 2, 3, 4, 5, 6, and 10 hours post "time zero" at Weeks 4, 8, 16, and 24
Population: Participants in the RTV PK Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | TVD + ATV/r + Iohexol | ABC/3TC + ATV/r + Iohexol
Number analyzed (Participants) | 16 | 17
hours
  Week 4 | 24.0 [24.0 to 24.0] | 24.0 [24.0 to 24.0]
  Week 8 | 24.0 [24.0 to 24.0] | 24.0 [24.0 to 24.0]
  Week 16: number analyzed (Participants) | 15 | 17
  Week 16 | 24.0 [24.0 to 24.0] | 24.0 [24.0 to 24.0]
  Week 24: number analyzed (Participants) | 15 | 17
  Week 24 | 24.0 [24.0 to 24.0] | 24.0 [24.0 to 24.0]

22. Secondary Outcome: PK Parameter: Ctau for RTV
Time Frame: Pre-dose, 0, 0.5, 1, 2, 3, 4, 5, 6, and 10 hours post "time zero" at Weeks 4, 8, 16, and 24
Population: Participants in the RTV PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TVD + ATV/r + Iohexol | ABC/3TC + ATV/r + Iohexol
Number analyzed (Participants) | 16 | 17
ng/mL
  Week 4 | 59.5 (57.85) | 61.0 (56.51)
  Week 8 | 71.0 (91.24) | 85.5 (99.68)
  Week 16: number analyzed (Participants) | 15 | 17
  Week 16 | 69.2 (49.85) | 99.1 (92.42)
  Week 24: number analyzed (Participants) | 15 | 17
  Week 24 | 102.5 (182.16) | 157.0 (246.75)

23. Secondary Outcome: PK Parameter: AUCtau for RTV
Time Frame: Pre-dose, 0, 0.5, 1, 2, 3, 4, 5, 6, and 10 hours post "time zero" at Weeks 4, 8, 16, and 24
Population: Participants in the RTV PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | TVD + ATV/r + Iohexol | ABC/3TC + ATV/r + Iohexol
Number analyzed (Participants) | 16 | 17
h*ng/mL
  Week 4 | 8259.6 (3166.47) | 9649.1 (3713.87)
  Week 8 | 8362.0 (3544.53) | 9702.2 (3391.68)
  Week 16: number analyzed (Participants) | 15 | 17
  Week 16 | 8102.6 (3392.00) | 11148.0 (4482.33)
  Week 24: number analyzed (Participants) | 15 | 16
  Week 24 | 8907.0 (5182.65) | 12039.3 (6792.06)

24. Secondary Outcome: PK Parameter: λz for RTV
Time Frame: Pre-dose, 0, 0.5, 1, 2, 3, 4, 5, 6, and 10 hours post "time zero" at Weeks 4, 8, 16, and 24
Population: Participants in the RTV PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | TVD + ATV/r + Iohexol | ABC/3TC + ATV/r + Iohexol
Number analyzed (Participants) | 16 | 17
1/hour
  Week 4: number analyzed (Participants) | 14 | 15
  Week 4 | 0.156 (0.0386) | 0.151 (0.0346)
  Week 8: number analyzed (Participants) | 13 | 15
  Week 8 | 0.144 (0.0474) | 0.142 (0.0281)
  Week 16: number analyzed (Participants) | 12 | 17
  Week 16 | 0.138 (0.0382) | 0.131 (0.0291)
  Week 24: number analyzed (Participants) | 15 | 15
  Week 24 | 0.133 (0.0347) | 0.128 (0.0469)

25. Secondary Outcome: PK Parameter: t1/2 for RTV
Time Frame: Pre-dose, 0, 0.5, 1, 2, 3, 4, 5, 6, and 10 hours post "time zero" at Weeks 4, 8, 16, and 24
Population: Participants in the RTV PK Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | TVD + ATV/r + Iohexol | ABC/3TC + ATV/r + Iohexol
Number analyzed (Participants) | 16 | 17
hours
  Week 4: number analyzed (Participants) | 14 | 15
  Week 4 | 4.56 [3.77 to 4.99] | 4.53 [3.83 to 6.01]
  Week 8: number analyzed (Participants) | 13 | 15
  Week 8 | 4.85 [3.75 to 5.34] | 4.68 [4.31 to 5.69]
  Week 16: number analyzed (Participants) | 12 | 17
  Week 16 | 5.39 [4.22 to 6.22] | 5.57 [4.68 to 6.00]
  Week 24: number analyzed (Participants) | 15 | 15
  Week 24 | 5.08 [4.49 to 5.78] | 4.82 [4.25 to 6.41]

26. Secondary Outcome: PK Parameter: Cmax for TFV
Time Frame: Pre-dose, 0, 0.5, 1, 2, 3, 4, 5, 6, and 10 hours post "time zero" at Weeks 4, 8, 16, and 24
Population: Participants in the TFV PK Analysis Set (all treated participants who have respective, evaluable PK profiles of TFV) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | STB + Iohexol | TVD + ATV/r + Iohexol | ATR + Iohexol
Number analyzed (Participants) | 17 | 16 | 15
ng/mL
  Week 4 | 371.2 (94.46) | 301.6 (116.36) | 298.3 (100.36)
  Week 8: number analyzed (Participants) | 17 | 16 | 14
  Week 8 | 379.8 (87.44) | 343.0 (133.97) | 325.5 (149.48)
  Week 16: number analyzed (Participants) | 17 | 15 | 15
  Week 16 | 399.5 (169.51) | 319.4 (146.41) | 298.6 (107.11)
  Week 24: number analyzed (Participants) | 16 | 15 | 15
  Week 24 | 394.4 (131.09) | 350.7 (126.91) | 305.9 (106.24)

27. Secondary Outcome: PK Parameter: Tmax for TFV
Time Frame: Pre-dose, 0, 0.5, 1, 2, 3, 4, 5, 6, and 10 hours post "time zero" at Weeks 4, 8, 16, and 24
Population: Participants in the TFV PK Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | STB + Iohexol | TVD + ATV/r + Iohexol | ATR + Iohexol
Number analyzed (Participants) | 17 | 16 | 15
hours
  Week 4 | 2.0 [1.3 to 3.1] | 3.0 [1.5 to 3.1] | 1.1 [0.6 to 2.0]
  Week 8: number analyzed (Participants) | 17 | 16 | 14
  Week 8 | 2.0 [2.0 to 2.1] | 3.0 [2.0 to 3.1] | 1.0 [0.6 to 1.1]
  Week 16: number analyzed (Participants) | 17 | 15 | 15
  Week 16 | 2.1 [1.1 to 3.1] | 2.1 [1.0 to 3.1] | 1.2 [1.0 to 2.1]
  Week 24: number analyzed (Participants) | 16 | 15 | 15
  Week 24 | 2.0 [1.1 to 3.0] | 2.1 [1.1 to 3.2] | 1.1 [0.6 to 2.0]

28. Secondary Outcome: PK Parameter: Clast for TFV
Time Frame: Pre-dose, 0, 0.5, 1, 2, 3, 4, 5, 6, and 10 hours post "time zero" at Weeks 4, 8, 16, and 24
Population: Participants in the TFV PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | STB + Iohexol | TVD + ATV/r + Iohexol | ATR + Iohexol
Number analyzed (Participants) | 17 | 16 | 15
ng/mL
  Week 4 | 81.1 (32.41) | 73.1 (23.74) | 55.4 (15.52)
  Week 8: number analyzed (Participants) | 17 | 16 | 14
  Week 8 | 80.9 (35.12) | 78.2 (31.27) | 53.4 (18.83)
  Week 16: number analyzed (Participants) | 17 | 15 | 15
  Week 16 | 128.5 (184.17) | 74.5 (26.01) | 63.0 (19.25)
  Week 24: number analyzed (Participants) | 16 | 15 | 15
  Week 24 | 78.5 (53.04) | 87.3 (41.20) | 58.5 (16.45)

29. Secondary Outcome: PK Parameter: Tlast for TFV
Description: as for outcome 21
Time Frame: Pre-dose, 0, 0.5, 1, 2, 3, 4, 5, 6, and 10 hours post "time zero" at Weeks 4, 8, 16, and 24
Population: Participants in the TFV PK Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | STB + Iohexol | TVD + ATV/r + Iohexol | ATR + Iohexol
Number analyzed (Participants) | 17 | 16 | 15
hours
  Week 4 | 24.0 [24.0 to 24.0] | 24.0 [24.0 to 24.0] | 24.0 [24.0 to 24.0]
  Week 8: number analyzed (Participants) | 17 | 16 | 14
  Week 8 | 24.0 [24.0 to 24.0] | 24.0 [24.0 to 24.0] | 24.0 [24.0 to 24.0]
  Week 16: number analyzed (Participants) | 17 | 15 | 15
  Week 16 | 24.0 [24.0 to 24.0] | 24.0 [24.0 to 24.0] | 24.0 [24.0 to 24.0]
  Week 24: number analyzed (Participants) | 16 | 15 | 15
  Week 24 | 24.0 [24.0 to 24.0] | 24.0 [24.0 to 24.0] | 24.0 [24.0 to 24.0]

30. Secondary Outcome: PK Parameter: Ctau for TFV
Time Frame: Pre-dose, 0, 0.5, 1, 2, 3, 4, 5, 6, and 10 hours post "time zero" at Weeks 4, 8, 16, and 24
Population: Participants in the TFV PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | STB + Iohexol | TVD + ATV/r + Iohexol | ATR + Iohexol
Number analyzed (Participants) | 17 | 16 | 15
ng/mL
  Week 4 | 74.6 (36.88) | 73.1 (23.74) | 55.4 (15.52)
  Week 8: number analyzed (Participants) | 17 | 16 | 14
  Week 8 | 75.8 (40.16) | 78.2 (31.27) | 48.8 (23.27)
  Week 16: number analyzed (Participants) | 17 | 15 | 15
  Week 16 | 128.5 (184.17) | 74.5 (26.01) | 57.5 (24.41)
  Week 24: number analyzed (Participants) | 17 | 15 | 15
  Week 24 | 71.7 (57.06) | 77.3 (43.06) | 54.2 (22.17)

31. Secondary Outcome: PK Parameter: λz for TFV
Time Frame: Pre-dose, 0, 0.5, 1, 2, 3, 4, 5, 6, and 10 hours post "time zero" at Weeks 4, 8, 16, and 24
Population: Participants in the TFV PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | STB + Iohexol | TVD + ATV/r + Iohexol | ATR + Iohexol
Number analyzed (Participants) | 17 | 16 | 15
1/hour
  Week 4: number analyzed (Participants) | 17 | 15 | 15
  Week 4 | 0.045 (0.0148) | 0.048 (0.0059) | 0.037 (0.0133)
  Week 8: number analyzed (Participants) | 17 | 15 | 13
  Week 8 | 0.051 (0.0167) | 0.048 (0.0158) | 0.041 (0.0197)
  Week 16: number analyzed (Participants) | 16 | 14 | 15
  Week 16 | 0.047 (0.0173) | 0.047 (0.0115) | 0.033 (0.0166)
  Week 24: number analyzed (Participants) | 16 | 15 | 15
  Week 24 | 0.051 (0.0195) | 0.046 (0.0184) | 0.035 (0.0138)

32. Secondary Outcome: PK Parameter: AUCtau for TFV
Time Frame: Pre-dose, 0, 0.5, 1, 2, 3, 4, 5, 6, and 10 hours post "time zero" at Weeks 4, 8, 16, and 24
Population: Participants in the TFV PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | STB + Iohexol | TVD + ATV/r + Iohexol | ATR + Iohexol
Number analyzed (Participants) | 17 | 16 | 15
h*ng/mL
  Week 4 | 3370.2 (1000.75) | 3151.2 (1107.18) | 2244.8 (572.09)
  Week 8: number analyzed (Participants) | 17 | 16 | 14
  Week 8 | 3549.7 (1238.03) | 3361.9 (1152.04) | 2250.8 (555.79)
  Week 16: number analyzed (Participants) | 17 | 15 | 15
  Week 16 | 3939.7 (2499.63) | 3234.7 (1207.58) | 2326.4 (494.24)
  Week 24: number analyzed (Participants) | 16 | 15 | 15
  Week 24 | 3307.0 (1387.97) | 3451.5 (1075.47) | 2265.7 (412.87)

33. Secondary Outcome: PK Parameter: t1/2 for TFV
Time Frame: Pre-dose, 0, 0.5, 1, 2, 3, 4, 5, 6, and 10 hours post "time zero" at Weeks 4, 8, 16, and 24
Population: Participants in the TFV PK Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | STB + Iohexol | TVD + ATV/r + Iohexol | ATR + Iohexol
Number analyzed (Participants) | 17 | 16 | 15
hours
  Week 4: number analyzed (Participants) | 17 | 15 | 15
  Week 4 | 15.73 [12.49 to 18.90] | 14.10 [13.28 to 16.81] | 20.65 [15.30 to 26.75]
  Week 8: number analyzed (Participants) | 17 | 16 | 13
  Week 8 | 14.40 [12.07 to 16.83] | 15.82 [11.94 to 19.53] | 18.81 [13.08 to 25.14]
  Week 16: number analyzed (Participants) | 16 | 14 | 15
  Week 16 | 14.41 [13.11 to 19.87] | 14.72 [12.76 to 16.73] | 22.78 [16.88 to 32.15]
  Week 24: number analyzed (Participants) | 16 | 15 | 15
  Week 24 | 13.99 [11.91 to 18.52] | 16.17 [13.18 to 21.37] | 21.54 [19.39 to 27.32]

34. Secondary Outcome: PK Parameter: AUCinf for Iohexol
Description: AUC inf is defined as the concentration of drug extrapolated to infinite time (area under the plasma concentration versus time curve extrapolated to infinite time).
Time Frame: Pre-dose, 0, 0.5, 1, 2, 3, 4, 5, 6, and 10 hours post "time zero" on Day 1 and Weeks 4, 8, 16, and 24
Population: Participants in the iohexol PK Analysis Set (all treated participants who have respective, evaluable PK profiles of iohexol) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*µg/mL
Groups:
- ATR + Iohexol: ATR (600/200/300 mg) FDC tablet orally once daily on an empty stomach for 24 weeks + iohexol 1500 mg solution administered intravenously at Baseline (Day 1), and Weeks 4, 8, 16, and 24
Arm/Group | STB + Iohexol | TVD + ATV/r + Iohexol | ATR + Iohexol | ABC/3TC + ATV/r + Iohexol
Number analyzed (Participants) | 17 | 16 | 16 | 17
h*µg/mL
  Day 1 | 511.2 (172.71) | 486.8 (108.28) | 706.9 (647.25) | 695.2 (523.33)
  Week 4: number analyzed (Participants) | 17 | 16 | 14 | 17
  Week 4 | 521.8 (121.67) | 496.2 (153.05) | 512.6 (163.89) | 720.5 (657.95)
  Week 8: number analyzed (Participants) | 17 | 16 | 15 | 16
  Week 8 | 517.8 (170.24) | 574.8 (382.63) | 510.6 (136.40) | 667.0 (559.06)
  Week 16: number analyzed (Participants) | 17 | 15 | 15 | 17
  Week 16 | 494.3 (113.60) | 509.5 (156.98) | 504.8 (95.07) | 725.9 (843.22)
  Week 24: number analyzed (Participants) | 17 | 15 | 15 | 17
  Week 24 | 545.8 (127.34) | 561.2 (214.26) | 507.1 (113.45) | 606.5 (321.40)

35. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL Week 24 as Determined by Snapshot Algorithm
Time Frame: Week 24
Population: Full Analysis Set (FAS): all participants who (1) are randomized into the study and (2) have received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | STB + Iohexol | TVD + ATV/r + Iohexol | ATR + Iohexol | ABC/3TC + ATV/r + Iohexol
Number analyzed (Participants) | 17 | 16 | 13 | 15
percentage of participants | 88.2 | 81.3 | 81.3 | 88.2

36. Secondary Outcome: Change From Baseline in Cluster of Differentiation 4 Positive (CD4+) Cell Count at Week 24
Time Frame: Baseline; Week 24
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | STB + Iohexol | TVD + ATV/r + Iohexol | ATR + Iohexol | ABC/3TC + ATV/r + Iohexol
Number analyzed (Participants) | 16 | 15 | 15 | 17
cells/uL | 139.63 (142.196) | 217.60 (195.375) | 204.33 (194.653) | 237.29 (201.222)

37. Secondary Outcome: Percentage of Participants Experiencing Adverse Events (AEs)
Description: Incidences of adverse events and laboratory abnormalities will be summarized.
Time Frame: Up to the last dose date plus 30 days (Up to 24 weeks plus 30 days)
Population: Safety Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | STB + Iohexol | TVD + ATV/r + Iohexol | ATR + Iohexol | ABC/3TC + ATV/r + Iohexol
Number analyzed (Participants) | 17 | 16 | 16 | 17
Percentage of participants
  Any Treatment-Emergent Adverse Events (TEAE) | 70.6 | 87.5 | 87.5 | 88.2
  Any Grade 3 or 4 Treatment-Emergent Adverse Event | 5.9 | 12.5 | 12.5 | 5.9
  Any Treatment-Emergent Study-Drug-Related AEs | 11.8 | 50.0 | 68.8 | 23.5
  Any TEAE Leading to Study Drug Discontinuation | 5.9 | 6.3 | 6.3 | 0

38. Secondary Outcome: Percentage of Participants Experiencing Treatment Emergent (TE) Grade 3 or 4 Laboratory Abnormalities
Description: Graded laboratory abnormalities were defined as values that increased at least one toxicity grade from predose at any postdose up to the last dose date of study drug plus 30 days. The most severe graded abnormality from all tests was counted for each participant.
Time Frame: Up to the last dose date plus 30 days (Up to 24 weeks plus 30 days)
Population: Safety Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | STB + Iohexol | TVD + ATV/r + Iohexol | ATR + Iohexol | ABC/3TC + ATV/r + Iohexol
Number analyzed (Participants) | 17 | 16 | 16 | 17
Percentage of participants
  Any Grade 3 or 4 TE Laboratory Abnormality | 5.9 | 25.0 | 12.5 | 52.9
  Grade 3 or 4 Neutrophils | 0 | 6.3 | 0 | 0
  Grade 3 or 4 Amylase | 0 | 0 | 6.3 | 0
  Grade 3 or 4 AST | 0 | 6.3 | 0 | 0
  Grade 3 or 4 CK | 5.9 | 18.8 | 6.3 | 5.9
  Grade 3 or 4 Total Bilirubin | 0 | 12.5 | 0 | 52.9
  Grade 3 or 4 Urine RBC | 0 | 7.7 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to 30 days after last dose of study drug (up to 24 weeks plus 30 days)
Description: Safety Analysis Set
Arm/Group | STB + Iohexol | TVD + ATV/r + Iohexol | ATR + Iohexol | ABC/3TC + ATV/r + Iohexol
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16 | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 1/17 | 1/16 | 1/16 | 2/17
Other Adverse Events (participants affected / at risk) | 11/17 | 14/16 | 13/16 | 14/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | STB + Iohexol (N=17) | TVD + ATV/r + Iohexol (N=16) | ATR + Iohexol (N=16) | ABC/3TC + ATV/r + Iohexol (N=17)
LIVER INJURY (Hepatobiliary disorders) | 0 | 1 | 0 | 0
ANAL ABSCESS (Infections and infestations) | 0 | 0 | 0 | 1
PNEUMONIA BACTERIAL (Infections and infestations) | 0 | 0 | 1 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
INTENTIONAL SELF-INJURY (Psychiatric disorders) | 0 | 0 | 0 | 1
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | STB + Iohexol (N=17) | TVD + ATV/r + Iohexol (N=16) | ATR + Iohexol (N=16) | ABC/3TC + ATV/r + Iohexol (N=17)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
EYE PAIN (Eye disorders) | 1 | 0 | 0 | 0
OCULAR ICTERUS (Eye disorders) | 0 | 3 | 0 | 1
ANAL FISSURE (Gastrointestinal disorders) | 1 | 0 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 0 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 3 | 5 | 2 | 4
DIARRHOEA HAEMORRHAGIC (Gastrointestinal disorders) | 0 | 0 | 0 | 1
DRY MOUTH (Gastrointestinal disorders) | 1 | 0 | 0 | 0
DYSPEPSIA (Gastrointestinal disorders) | 0 | 1 | 0 | 1
FLATULENCE (Gastrointestinal disorders) | 1 | 0 | 0 | 1
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 2 | 0 | 1
TOOTHACHE (Gastrointestinal disorders) | 0 | 0 | 2 | 1
VOMITING (Gastrointestinal disorders) | 0 | 0 | 1 | 0
ASTHENIA (General disorders) | 0 | 0 | 0 | 1
FATIGUE (General disorders) | 2 | 1 | 0 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 1 | 1 | 1
PAIN (General disorders) | 0 | 0 | 1 | 0
PYREXIA (General disorders) | 0 | 1 | 0 | 0
JAUNDICE (Hepatobiliary disorders) | 0 | 2 | 0 | 1
SEASONAL ALLERGY (Immune system disorders) | 0 | 0 | 0 | 1
ACUTE HEPATITIS C (Infections and infestations) | 0 | 0 | 1 | 0
ANAL CHLAMYDIA INFECTION (Infections and infestations) | 0 | 1 | 0 | 0
CYSTITIS (Infections and infestations) | 0 | 0 | 1 | 0
EAR INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
EYE ABSCESS (Infections and infestations) | 0 | 1 | 0 | 0
EYELID BOIL (Infections and infestations) | 0 | 0 | 0 | 1
FUNGAL SKIN INFECTION (Infections and infestations) | 0 | 0 | 1 | 0
FURUNCLE (Infections and infestations) | 1 | 0 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 0 | 1
GONORRHOEA (Infections and infestations) | 0 | 3 | 1 | 1
LARYNGITIS (Infections and infestations) | 0 | 0 | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 1 | 3 | 3 | 2
ONYCHOMYCOSIS (Infections and infestations) | 0 | 1 | 0 | 0
OTITIS EXTERNA (Infections and infestations) | 0 | 0 | 1 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 1 | 0 | 0
SYPHILIS (Infections and infestations) | 1 | 0 | 0 | 0
TINEA CRURIS (Infections and infestations) | 1 | 0 | 0 | 0
TINEA PEDIS (Infections and infestations) | 2 | 0 | 0 | 0
TINEA VERSICOLOUR (Infections and infestations) | 0 | 0 | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0 | 1
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 | 2 | 0 | 0
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 | 1 | 0 | 0
INCREASED APPETITE (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
ANOGENITAL WARTS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
DIZZINESS (Nervous system disorders) | 0 | 1 | 7 | 0
HEAD DISCOMFORT (Nervous system disorders) | 0 | 1 | 0 | 0
HEADACHE (Nervous system disorders) | 2 | 1 | 2 | 3
HYPOAESTHESIA (Nervous system disorders) | 1 | 0 | 0 | 0
LETHARGY (Nervous system disorders) | 0 | 1 | 0 | 0
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 0 | 0 | 1 | 0
ABNORMAL BEHAVIOUR (Psychiatric disorders) | 0 | 1 | 0 | 0
ABNORMAL DREAMS (Psychiatric disorders) | 0 | 0 | 1 | 0
DEPRESSED MOOD (Psychiatric disorders) | 0 | 1 | 1 | 0
DISORIENTATION (Psychiatric disorders) | 1 | 0 | 0 | 0
INDIFFERENCE (Psychiatric disorders) | 1 | 0 | 0 | 0
INSOMNIA (Psychiatric disorders) | 1 | 0 | 1 | 2
NIGHTMARE (Psychiatric disorders) | 0 | 0 | 2 | 0
SLEEP DISORDER (Psychiatric disorders) | 1 | 0 | 0 | 0
TERMINAL INSOMNIA (Psychiatric disorders) | 0 | 1 | 0 | 0
CATARRH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 0
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
HAEMATOMA (Vascular disorders) | 1 | 0 | 1 | 0
HOT FLUSH (Vascular disorders) | 0 | 0 | 1 | 0
HYPOTENSION (Vascular disorders) | 0 | 1 | 0 | 0
SPIDER VEIN (Vascular disorders) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
There were no limitations affecting the analysis or results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years